CLINICAL TRIAL: NCT00652782
Title: A Randomized, Double-Blind, Placebo Controlled Dose-Ranging Study of The Effects of MK7418, Both as Monotherapy and in Combination With Furosemide, On Diuresis and Renal Function in Patients With Congestive Heart Failure (CHF) And Renal Impairment Treated With Oral Loop Diuretics Who Require Hospitalization For Fluid Overload
Brief Title: Effects of MK7418 on Diuresis and Renal Function in Congestive Heart Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaCardia, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007_806; MK7418-201
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: Congestive Heart Failure; Renal Impairment
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — rolofylline

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): rolofyline 2.5 mg IV QD
  Interventions: Drug: rolofyline
- 2 (Experimental): rolofyline 15 mg IV QD
  Interventions: Drug: rolofyline
- 3 (Experimental): rolofyline 30 mg IV QD
  Interventions: Drug: rolofyline
- 4 (Experimental): rolofyline 60 mg IV QD
  Interventions: Drug: rolofyline
- 5 (Placebo Comparator): placebo for rolofyline IV QD
  Interventions: Drug: Comparator Placebo (unspecified)

INTERVENTIONS:
Drug: rolofyline — rolofyline 2.5 mg IV QD; 15 mg IV QD; 30 mg IV QD; 60 mg IV QD; 3 days
  Other Names: MK7418
  Arms: 1; 2; 3; 4
Drug: Comparator Placebo (unspecified) — Matching placebo for rolofyline IV QD; 3 days
  Arms: 5

SUMMARY:
A study to determine the most appropriate dose of MK7418 in heart failure patients presenting with symptoms of volume overload requiring increased diuretic doses.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide written informed consent,
* Be a male or female at least 18 years of age,
* Be hospitalized for fluid overload requiring IV diuretic therapy
* History of use of diuretic therapy for CHF (including this admission),
* Be admitted to the hospital within 36 hours of the mandatory dose of IV furosemide 40 mg at between 2000 and 2200 hour on Day -1

Exclusion Criteria:

* Have had a myocardial infarction within 30 days prior to Day -1
* Be pregnant or breast-feeding
* Have received intravascular contrast material within the preceding 14 days; or have acute contrast nephropathy
* Have had implantation of an automated implanted cardiac defibrillator (AICD) or synchronization device within the preceding 7 days
* Currently require mechanical ventilation, ultrafiltration, or hemodialysis,
* Have symptomatic ventricular tachycardia
* Be admitted for heart transplant surgery or have had a heart transplant,
* Have any other concomitant life-threatening disease,
* Have participated in a clinical trial of an investigational drug or device within 30 days before randomization
* Have a positive urine pregnancy test (for women of child-bearing capacity)
* Have an allergy to soybean oil and/or eggs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-12; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To measure the diuretic effect of a single dose of the study medication (monotherapy) over six hours compared to a single dose of IV placebo (monotherapy) in CHF patients with renal impairment | 30 days

SECONDARY OUTCOMES:
To determine the optimal dose range of intravenous (IV) study medication combination with IV furosemide, with or without other diuretics, in preventing deterioration of renal function in CHF patients | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC